CLINICAL TRIAL: NCT05767853
Title: Multiparametric Assessment of Peripheral Blood and Tissue Myeloid Cells Phenotype Associated With Severe Lung Manifestations and Cytokines Storm for Precision Medicine in Patients With SARS-Cov-2 Infection.
Brief Title: Multiparametric Assessment of Peripheral Blood and Tissue Myeloid Cells. Phenotype for Precision Medicine in Patients With SARS-Cov-2 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Alivernini Stefano, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3213
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Pneumonia
Keywords: bronchoalveolar lavage fluid; peripheral blood

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-Cov-2pos pneumonia with moderate/severe lung manifestations with clinical worsening: (PaO2/FiO2<200)
  Interventions: Other: Immune-phenotyping of tissue and peripheral blood myeloid compartment
- SARS-Cov-2pos pneumonia with moderate/severe lung manifestations with clinical improvement: (PaO2/FiO2>200)
  Interventions: Other: Immune-phenotyping of tissue and peripheral blood myeloid compartment

INTERVENTIONS:
Other: Immune-phenotyping of tissue and peripheral blood myeloid compartment — Peripheral blood sampling and bronchoalveolar lavage fluid collection based on the clinical indication at baseline (T0) and peripheral blood sample at the time of clinical worsening/improvement during the follow-up (T1). Moreover, after complete recovery and discharge from the hospital peripheral blood sampling in the outpatient clinical assessment will be performed (T2).
  BALF and peripheral blood will be processed for immune-phenotyping of the myeloid compartment using single-cell RAN sequencing analysis.

SUMMARY:
We hypothesise that patients with SARS-Cov-2 infection are characterized by progressive changes in distribution of distinct lung macrophages populations mediated by influx of circulating monocytes into the lungs . Moreover, we also hypothesise that patients with higher rate of MerTKpos alveolar macrophages in the lung lavage will have the lowest rate of lung complications and the best recovery outcome in terms of clinical outcome and need of assisted ventilation supporting the use of macrophage phenotyping as novel prognostic biomarker in patients with SARS-Cov-2 infection. Finally, the definition of the transcriptomic signature of peripheral blood and tissue-derived myeloid cell subtypes will offer new therapeutic target of this uncurable newly discovered infection.

ELIGIBILITY:
Inclusion Criteria:

- Patients with COVID-19 pneumonia

Exclusion Criteria:

* Other infections rather than Covid-19
* Patients with concomitant treatment with prednisone ≥10 mg daily
* Patients under therapy with immunosuppressants

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospedalized for Covid-19 pneumonia.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement as shown by PaO2/FiO2>200 | 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- Division of Rheumatology, Rome, Lazio, Italy
- School of Infection and Immunity, Glasgow, United Kingdom